CLINICAL TRIAL: NCT02199535
Title: The Analysis of the Risks of the Personnel Working in Anesthesiology Departments in Turkey
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Günay CANPOLAT, assoc. Prof, TC Erciyes University
Other Study IDs: 2014/340
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Exposure
Keywords: operating room,; risk factors; anesthesiologists

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study was to investigate the analysis of the risks faced by the personnel working in the field of Anesthesiology and Reanimation in Turkey

DETAILED DESCRIPTION:
There are many potential risks in operating room such as anesthetic gas exposure, chronic noise, fair, intensive working conditions, frequent guardians of the doctors and anesthesia staff. Those are effects the staff of anesthesia such as doctors, anesthesia assistants, anesthesia nurses. They usually suffer from hard working, fatigue and exposing anesthetic gases effects them as well. These reasons cause some undesirable adverse effects. The scientific dates are really limited in uour country. We aimed to ask questions the anesthesia staff and determine the environment conditions and the other risk in operating room that effects the staff. For t his purpose we prepared a questionaire and send to their e-mail address.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia doctors anesthesia nurses anesthesia technic personal

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The anesthesia staff doctors nurses and anesthesia personal
Sampling Method: Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The analysis of the risks in the operating room | during 1 months
  This a questionnaire study. We prepared a questionnaire and send it to anesthesia staff by e-mail address. their reply will evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)